CLINICAL TRIAL: NCT06467721
Title: Clinical Efficacy of Self-adhesive Silicone Gel Waterproof Dressings Versus Conventional Dressings in the Healing of Incisions After Total Joint Arthroplasty: a Prospective, Randomized Controlled Trial Study
Brief Title: Clinical Efficacy of Self-adhesive Silicone Gel Waterproof Dressings Versus Conventional Dressings in the Healing of Incisions After Total Joint Arthroplasty
Acronym: Yes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Long Hua, Principal Investigator, First Affiliated Hospital of Xinjiang Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: XJ202405-01
Record Dates: First submitted 2024-06-10; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Self-adhesive Silicone Gel Waterproof Dressing; Gauze Dressing; Total Joint Arthroplasty
Keywords: self-adhesive silicone gel waterproof dressing; gauze dressing; total joint arthroplasty; RCT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-adhesive silicone gel waterproof dressing group (Experimental): Self-adhesive silicone gel waterproof dressing is used after artificial joint replacement surgery
  Interventions: Device: Self-adhesive silicone gel waterproof dressing
- Sterile gauze dressing group (Active Comparator): Sterile gauze dressing is used after artificial joint replacement surgery
  Interventions: Device: Sterile gauze dressing

INTERVENTIONS:
Device: Self-adhesive silicone gel waterproof dressing — Self-adhesive silicone gel waterproof dressing is used after artificial joint replacement surgery.
  Arms: Self-adhesive silicone gel waterproof dressing group
Device: Sterile gauze dressing — Sterile gauze dressing is used after artificial joint replacement surgery.
  Arms: Sterile gauze dressing group

SUMMARY:
The efficacy of using self-adhesive silicone gel waterproof dressings versus conventional gauze dressings for recovery after total joint arthroplasty (TJA) remains unclear. In our study, we conducted a prospective, randomized controlled trial to compare these two types of dressings. Patients were divided into two groups following TJA, and we collected primary outcome measures such as skin infection rate and re-operation rate. Additionally, we gathered blood inflammatory indicators, including C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR), to evaluate the effectiveness of the two treatments. Finally, we perform one year follow up including REEDA score, MSS score to evaluate the recovery of the skin.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender is not limited;
2. Meet the diagnostic criteria for artificial joint replacement;
3. Initial joint replacement surgery;
4. Voluntary and signed informed consent.

Exclusion Criteria:

1. Allergic to self-adhesive silicone rubber waterproof dressing;
2. Patients with severe knee joint infection who cannot undergo artificial joint replacement;
3. Progressive renal insufficiency (stage 4 and above) or glomerular filtration rate less than 30ml/min;
4. periprosthesis infection after multiple joint replacement;
5. Active infection at the site of intravenous or joint injection;
6. long-term use of anticoagulants or antiplatelet drugs due to other diseases;
7. Have sepsis or positive blood culture within the last 30 days;
8. Radiotherapy and chemotherapy are required due to neoplastic diseases;
9. Receiving systemic glucocorticoid therapy (prednisone > 10mg/ day or equivalent hormone medication);
10. severe immunodeficiency diseases (such as stage 3 HIV, sickle cell anemia, splenectomy, etc.);
11. Have a history of drug abuse;
12. Treatment of bone marrow or other transplants with immunosuppressive drugs;
13. Pregnant, parturient and lactating women;
14. Participating in other clinical trials;
15. Researchers believe that other reasons are not appropriate for clinical trial participants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Infection control rate | One month and three month after surgery
  Calculate the infection control rate in the two groups
Redness, Edema, Ecchymosis, Discharge, and Approximation score (REEDA score) | One day before surgery, three month after surgery
  The REEDA score is a clinical tool used to assess the healing of perineal wounds and other skin wounds, particularly after childbirth. REEDA stands for Redness, Edema, Ecchymosis, Discharge, and Approximation. Each of these five parameters is scored on a scale from 0 to 3, with higher scores indicating more severe symptoms. The total REEDA score can range from 0 to 15.
Modified Severity Score (MSS) | One day before surgery, three month after surgery
  This score is often used in dermatology to evaluate the severity of conditions such as atopic dermatitis or other chronic skin disorders. The MSS score helps clinicians to quantify the extent and severity of skin involvement, aiding in treatment decisions and monitoring progress.

SECONDARY OUTCOMES:
X-ray | One day before surgery and three months after surgery.
  X-ray of surgery site.
American Knee Society Score (AKS score) | One day before surgery and three months after surgery.
  American Knee Society Score is used to evaluate the outcomes of knee replacement surgery. This scoring system consists of two main components: the knee score and the function score.
The Harris Hip Score (HHS) | One day before surgery and three months after surgery.
  The Harris Hip Score (HHS) is a widely used clinical tool for assessing the outcomes of hip surgeries, particularly hip replacements. Developed by Dr. William Harris in 1969, it evaluates various aspects of hip function and pain to provide an overall score that reflects the patient's condition. The higher the score, the better the result is.
Visual Analog Scale (VAS score) | One day before surgery and three months after surgery.
  The VAS score, or Visual Analog Scale, is a tool commonly used to measure a person's level of pain. The VAS is a simple, subjective measure that consists of a straight line, typically 10 centimeters long, anchored by two endpoints. One end of the line represents "no pain" and the other end represents "worst pain imaginable." For example, if the VAS line is 10 cm long and the patient's mark is at 7 cm from the "no pain" end, their pain score would be 7 out of 10.
Alanine Aminotransferase (ALT) | One day before surgery and one day after surgery
  An enzyme found in the liver that helps convert proteins into energy. Elevated levels indicate liver damage. Normal range: 10 to 40 units per liter (U/L)
Aspartate Aminotransferase (AST) | One day before surgery and one day after surgery
  An enzyme found in the liver and other tissues. High levels can indicate liver damage but are less specific than ALT. Normal range: 10 to 40 units per liter (U/L)
Serum Creatinine | One day before surgery and one day after surgery
  Measures the level of creatinine in the blood. Elevated levels can indicate impaired kidney function. Normal range: 62 to 115 micromoles per liter (µmol/L).
Blood Urea Nitrogen （BUN） | One day before surgery and one day after surgery
  Measures the amount of nitrogen in the blood that comes from urea. Elevated BUN levels can indicate impaired kidney function. Normal range: 2.5 to 7.1 millimoles per liter (mmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Li Cao, Study Chair — The first affliated hospital, Xinjiang medical university

IPD SHARING:
Plan to Share IPD: Yes
Other researchers can contact the corresponding author after the research publishing.
Supporting Information: Study Protocol
Time Frame: Other researchers can contact the corresponding author after the research publishing.